CLINICAL TRIAL: NCT03666013
Title: Mitochondrial Health and Muscle Function in Elderly
Brief Title: Mitochondria and Muscle Health in Elderly
Acronym: ELMIH
Status: Completed | Type: Observational
Sponsor: Maastricht University (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government); Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Other Study IDs: Mitohealth
Record Dates: First submitted 2018-09-04; First posted 2018-09-11 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Muscle Weakness
Keywords: Mitochondrial health; Muscle function; Aging
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine, blood, muscle tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Young healthy subjects: 20-30 years old, max 1h of exercise per week
- Elderly with a normal physical function: 65-80 years old, max 1h of exercise per week
- Elderly with a decreased physical function: 65-80 years old, max 1h of exercise per week, SPPB under 9 or frailty score lower then 10
- Active elderly: 65-80 years old, minimal 3h of exercise per week

SUMMARY:
The aim of this study is to characterize the relation between skeletal muscle mitochondrial metabolism and muscle health in elderly, physically compromised humans. To study this relation, a cross-sectional study will be performed in well-defined, distinct subject groups. Thus, to obtain insight in the relation between mitochondrial health and muscle function, not only subjects that differ in mitochondrial function (based on physical activity) will be compared but also subjects with high- versus low muscle function will be selected.

DETAILED DESCRIPTION:
Aging is associated with a decline of mitochondrial and skeletal muscle volume, -quality and -function. If a causal link exists between the loss of mitochondrial function and muscle health is unknown, however, both appear with advancing age and are associated with the loss of functional capacity, which increases comorbidities and annual healthcare costs. The aim is to test the hypothesis that a compromised muscle function in sedentary elderly is related to an impaired mitochondrial health. A detailed characterization of mitochondrial metabolism and muscle function is performed in well-defined, (physically compromised) elderly humans, in a cross-sectional design. To obtain insight in the relation between mitochondrial health and muscle function, not only elderly subjects that differ in mitochondrial function (based on physical activity) will be compared but also elderly subjects with high versus low muscle physical function will be selected. Healthy, young (20-30 years,) individuals with normal physical activity levels will be included as absolute controls.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Subject should be in sufficient health to participate in the experimentations, to be judged by the responsible MD based on the subject's medical history
* Caucasian origin (see study groups)

Exclusion Criteria:

* Any contraindications for MRI scan:

Aneurysm clips Implanted neural stimulator Implanted cardiac pacemaker of defibrillator Cochlear implant Iron- containing corpora aliena in the eye or brain Artificial (heart) valves which is contraindicated for MRS Claustrophobia

* Diagnosed with diabetes mellitus
* Poor health as judged by the responsible medical doctor
* Heart problems: In case of an abnormal ECG in rest, this will be discussed with both the participant and the responsible medical doctor

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy volunteers between 20 and 30 years old and 65 and 80 years old
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Rate of ex vivo mitochondrial State 3 respiration | Day 4
  Ex vivo mitochondrial capacity, ADP-stimulated respiration expressed by O2flux in pmol/mg wet weight/second

SECONDARY OUTCOMES:
Insuline sensitivity | Day 1
  Measured by 1-step hyperinsulinemic euglycemic. Insulin-stimulated glucose disposal, expressed as the rate of disappearance of the glucose (Rd glucose in μmol*kg-1*bw*min-1
Physical functionality, 6MWT | Day 2
  Measured by a standardized 6-minute walk test. Physical functionality expressed in the distance (in meters) the subject is able to walk over a total of six minutes
VO2max | Day 2
  Maximal oxygen uptake measured by maximal cycling test (ml*kg-1*min-1)
Body composition | Day 3
  Measured by BodPod and expressed by percentages of fat mass (%)
Dynamic gait stability | Day 3
  Characterized by using the CAREN-system locomotion assessment and expressed by amount of steps necessary to regain normal walking pattern
Muscle strength in upper-leg | Day 3
  Extensor and flexor muscles of the knee joint measured by dynamometer (Biodex) expressed in peak torque 70° extension and flexion knee (Nm/kg)
Energy expenditure in rest and during sub-maximal exercise | Day 4
  indirect calorimetry during 45 minutes in resting state (in KJ/min) and 1-hour exercise bout at 50% of maximal power output (in KJ/min)
Muscle oxidative capacity in vivo (PCr-MRS recovery) | Day 5
  In vivo skeletal muscle PCr-recovery expressed by PCr halftime (s)
Muscle metabolism in vivo (H-MRS acetylcarnitine) | Day 5
  In vivo skeletal muscle acetylcarnitine concentrations in rest measured by H-MRS and expressed by mmol/kgww
Muscle volume upper-leg | Day 5
  Muscle volume measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, Prof . dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Mevenkamp J, Bruls YMH, Mancilla R, Grevendonk L, Wildberger JE, Brouwers K, Hesselink MKC, Schrauwen P, Hoeks J, Houtkooper RH, Buitinga M, de Graaf RA, Lindeboom L, Schrauwen-Hinderling VB. Development of a 31P magnetic resonance spectroscopy technique to quantify NADH and NAD+ at 3 T. Nat Commun. 2024 Oct 24;15(1):9159. doi: 10.1038/s41467-024-53292-4. PMID 39443469
- [Derived] Mancilla R, Pava-Mejia D, van Polanen N, de Wit V, Bergman M, Grevendonk L, Jorgensen J, Kornips E, Hoeks J, Hesselink MKC, Schrauwen-Hinderling VB. Invasive and noninvasive markers of human skeletal muscle mitochondrial function. Physiol Rep. 2023 Jun;11(12):e15734. doi: 10.14814/phy2.15734. PMID 37340318
- [Derived] Mancilla RF, Lindeboom L, Grevendonk L, Hoeks J, Koves TR, Muoio DM, Schrauwen P, Schrauwen-Hinderling V, Hesselink MK. Skeletal muscle mitochondrial inertia is associated with carnitine acetyltransferase activity and physical function in humans. JCI Insight. 2023 Jan 10;8(1):e163855. doi: 10.1172/jci.insight.163855. PMID 36413408